CLINICAL TRIAL: NCT07289880
Title: Efficacy of Diacylglycerol Oil on Metabolic Risk Factors in Prediabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Responsible Party: Principal Investigator, Qiu-ye Lan, Associate Researcher, Guangdong Pharmaceutical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FirstAHGuangdong
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Diglycerides

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAG Oil Group (Experimental): A four-week dietary intervention will be implemented, during which participants assigned to the intervention group will replace their habitual cooking oil with diacylglycerol (DAG) oil.
  Interventions: Combination Product: Diacylglycerol oil
- Control Group (Active Comparator): Participants assigned to the control group will consume colza oil as their cooking oil throughout a four-week dietary intervention. No other lifestyle habits or dietary behaviors will be altered.
  Interventions: Combination Product: Colza Oil

INTERVENTIONS:
Combination Product: Diacylglycerol oil — This study will implement a four-week dietary intervention in which participants assigned to the intervention group will replace their habitual cooking oil with diacylglycerol (DAG) oil. All other lifestyle behaviors will be maintained without modification.
  Arms: DAG Oil Group
Combination Product: Colza Oil — Participants assigned to the control group will consume colza oil as their cooking oil throughout a four-week dietary intervention. No other lifestyle habits or dietary behaviors will be altered.
  Arms: Control Group

SUMMARY:
This study will implement a four-week dietary intervention among middle-aged and older adults with pre-diabetes. Participants assigned to the intervention arm will replace their usual cooking oil with diacylglycerol (DAG) oil, while those in the control arm will consume colza oil. All other lifestyle behaviors will be maintained without modification. The trial will determine the impact of DAG oil consumption on glycemic regulation, lipid metabolism, and body composition in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40-75 years.
2. Diagnosed with prediabetes according to American Diabetes Association (ADA) criteria: including fasting plasma glucose (FPG) levels of 5.6-6.9 mmol/L, and/or 2-hour postprandial glucose (OGTT-2h) levels of 7.8-11.1 mmol/L, and/or glycated hemoglobin (HbA1c) levels of 5.7%-6.4%.
3. Body mass index (BMI) ≥ 24 kg/m².
4. No plans to relocate or travel extensively in the next three months.
5. Willing to consume all study-provided meals throughout the intervention.
6. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Diagnosis of diabetes (Type 1 or Type 2).
2. Current use of any glucose-lowering medication.
3. Use of appetite suppressants or hormonal medications.
4. History of bariatric surgery, or weight change >5% in the past 3 months.
5. Alcohol consumption >40 g/day.
6. Use of antibiotics, probiotics, or prebiotics within the past 3 months.
7. Pregnancy, lactation or planning pregnancy.
8. History of severe cardiovascular disease, malignancy, autoimmune disease, cognitive impairment, or severe dysfunction of thyroid, liver, kidney, or digestive system.
9. Inability to comprehend information, communicate effectively, or comply with the study protocol.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Continuous Glucose Monitoring (CGM) Data | up to 4 weeks
  At baseline, and 4 weeks, investigators will using Continuous Glucose Monitoring (CGM) to monitor the glucose level of participants.

SECONDARY OUTCOMES:
weight | up to 4 weeks
  At baseline, and 4 weeks, investigators will examine weight.
fasting blood glucose | At baseline and after 4 weeks of intervention
  At baseline, and 4 weeks, investigators will use automatic electrochemiluminescence analyzer to examine fasting blood glucose.
lipid metabolism | At baseline and after 4 weeks of intervention
  At baseline, and 4 weeks, investigators will use automatic electrochemiluminescence analyzer to examine total cholesterol, low density lipoprotein, high density lipoprotein, triglyceride.
HbA1c | At baseline and after 4 weeks of intervention
  At baseline, and 4 weeks, investigators will use automatic electrochemiluminescence analyzer to examine HbA1c.
intestinal bacteria | up to 4 weeks
  At baseline, and 4 weeks, investigators will use 16S rRNA pyrosequencing to examine intestinal bacteria.
TIR (time in range) | At baseline and after 4 weeks of intervention
  TIR refers to the time when blood glucose is controlled within a reasonable ( target ) range (3.9~10.0 mmol/L), measured by continuous glucose monitoring at baseline and 4 weeks.
sleep quality | up to 4 weeks
  Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI), which comprises seven components (A through G), each scored on a scale of 0-3. The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
blood pressure | up to 4 weeks
  At baseline, and 4 weeks, investigators will test the systolic blood pressure and diastolic blood pressure using automatic digital blood pressure monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Street, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No